CLINICAL TRIAL: NCT02199314
Title: The Effect of Anesthesia on the Recruitment of Motor Evoked Potentials Using an Increased Number of Pulses
Brief Title: Anesthesia and Motor Evoked Potential (MEP) Recruitment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2012-1065
Record Dates: First submitted 2014-04-11; First posted 2014-07-24 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2017-11

CONDITIONS: Idiopathic Scoliosis
Keywords: intra; operative; neurophysiologic; monitoring; transcranial; motor; evoked; potential; anesthesia; pulses
MeSH Terms: interventions — Desflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- desflurane MEP's (Experimental): Transcranial motor evoked potentials are obtained under total intravenous anesthesia (TIVA) and again after desflurane at 3%, for at least 5 minutes.at two different time points. Each subject is his/her own control
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Desflurane
  Other Names: Suprane

SUMMARY:
Test the hypothesis to recruit larger motor responses to transcranial stimulation.

DETAILED DESCRIPTION:
The study is designed to test the hypothesis that it is possible to recruit larger motor responses to transcranial stimulation by increasing the number of stimulating pulses under both baseline conditions and conditions of increased anesthetic suppression of the motor responses.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 through 17 years
* Diagnosis of idiopathic scoliosis
* Scheduled for posterior spinal fusion with neurophysiological monitoring
* No known allergies to propofol or remifentanil
* No contraindication to total intravenous anesthesia
* No contraindications to the administration of volatile agents

Exclusion Criteria:

* Failure to consent or assent to study
* Diagnosis other than idiopathic scoliosis
* Poorly controlled seizures or the presence of a cochlear implant
* Patient history or family history of malignant hypothermia or mitochondrial myopathies

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in Orthopaedics clinic during scheduled visit for pre-surgical planning. Parents/guardians were given the informed consent and participant were given assent documents. Anyone who agreed to participate at this time was considered enrolled for the purposes of the study. This number was 30.
Pre-assignment Details: There was no group assignment - each participant was to be his/her own control.
Groups:
- MEPs Pre and Post Desflurane at 2 Time Points: Transcranial motor evoked potentials are recorded under a TIVA anesthetic and again after addition of 3% desflurane for 5 minutes at two different time points in a surgical procedure
Period: Overall Study
Arm/Group | MEPs Pre and Post Desflurane at 2 Time Points
Started | 30
Completed | 14
Not Completed | 16
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 10

BASELINE CHARACTERISTICS:
Population: 30 participants initially enrolled. 12 were withrdrawn prior to any analysis. Data from 18 participants analyzed as 18 participants had part 1 of study procedures completed. 14 participants completed the study, that is had both part 1 and part 2 procedures.
Groups:
- Desflurane MEP's: Transcranial motor evoked potentials are obtained under propofol/remifentanil TIVA anesthesia and the again under TIVA plus desflurane 3%, after desflurane has been on for at least 5 minutes, at two different time points; before incision and at the end of the procedure. Each patient is his/her own control
Arm/Group | Desflurane MEP's
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] — Population: 30 participants initially enrolled. 12 were withdraw prior to start of study procedures. 6 withdrawn by participant and 6 by physician decision
  years | 14 [12 to 16]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: 30 participants initially enrolled. 12 were withdraw prior to start of study procedures. 6 withdrawn by participant and 6 by physician decision
  Participants
    Female | 14
    Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Effect of Pulse Train Length on Transcranial Motor Evoked Potentials (TcMEP) Area Under Total Intravenous Anesthesia (TIVA) and TIVA Plus 3% Desflurane
Description: A series of 15 transcranial motor evoked potentials are recorded under a TIVA anesthetic and again after addition of 3% desflurane for 5 minutes at two different time points in a surgical procedure. The series consisted of 3 runs of 5,6, 7, 8, and 9 pulse trains, each train separated by 30 seconds. The 3 runs were averaged to give and average value of TcMEP amplitude and area for the 5,6,7,8 and 9 pulse trains. The data were used to compute regression coefficients for area vs pulse length for the TIVA case and TIVA plus desflurane for each participant who completed the study..The final measure is the number of participants who had a MEP area ratios significantly different from 1 at all times and conditions; that is for TIVA alone and TIVA plus desflurane, at both time points.
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Groups:
- MEPs Pre and Post Desflurane at 2 Time Points: A series of 15 transcranial motor evoked potentials are recorded under a TIVA anesthetic and again after addition of 3% desflurane for 5 minutes at two different time points in a surgical procedure. The series consisted of 3 runs of 5,6, 7, 8, and 9 pulse trains, each train separated by 30 seconds. The 3 runs were averaged to give and average value of TcMEP amplitude and area for the 5,6,7,8 and 9 pulse trains. The data were used to compute regression coefficients for area vs pulse length for the TIVA case and TIVA plus desflurane for each participant who completed the study..
Arm/Group | MEPs Pre and Post Desflurane at 2 Time Points
Number analyzed (Participants) | 14
Participants | 2

ADVERSE EVENTS:
Groups:
- Desflurane MEP's: Transcranial motor evoked potentials are obtained under TIVA and again after desflurane at 3%, for at least 5 minutes.at two different time points. Each subject is his/her own control
  Desflurane
Arm/Group | Desflurane MEP's
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desflurane MEP's (N=18)
Enlarged thyroid (Endocrine disorders) | 1 (1) — Patient found to have enlarged thyroid gland at end of procedure - deemed unrelated to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes